CLINICAL TRIAL: NCT07187869
Title: Modulation of the Bone Immune Microenvironment Following Cabozantinib Treatment of Bone Metastatic Clear Cell Renal Cell Carcinoma: Proof of Concept Study
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0624; NCI-2025-06901 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-09-16; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Clear Cell Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — cabozantinib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with Cabozantinib [PO] + Nivolumab [IV] Q4W (Experimental): Participants standard of care treatment stage begins when the patient has completed the baseline paired core biopsies.
  Interventions: Drug: Cabozantinib; Drug: Nivolumab

INTERVENTIONS:
Drug: Cabozantinib — Given by IV
  Other Names: Cometriq; Cabometyx
Drug: Nivolumab — Given by IV
  Other Names: Opdivo

SUMMARY:
The goal of our study is to explore how treatments affect the bone immune microenvironment and determine the best treatment options for patients with metastatic kidney cancer to the bone. This could prevent skeletal complications and improve patient outcomes.

DETAILED DESCRIPTION:
Primary Objectives:

1. To assess safety of obtaining biopsy within close time frame of cabozantinib treatment.
2. To evaluate the success rate of obtaining serial biopsies of bone metastases. Success is defined as viable single cell sequencing of bone biopsy samples at baseline and after 8 weeks of treatment.
3. To quantify the fold change in M1:M2 macrophage population in serial biopsies from renal cell carcinoma bone metastases.

Secondary Objectives:

1. To compare the M1:M2 macrophage population at baseline and on therapy in paired bone versus non-bone metastatic sites.
2. To compare CD8+, Granzyme+ cells on multiplex immunofluorescence at baseline and on therapy in paired bone versus non-bone metastatic sites.
3. To describe serum marker changes over time while on therapy for bone metastasis including bone alkaline phosphatase, osteopontin, procollagen type I amino-terminal propeptide (PINP), and beta-isomer of carboxy-terminal telopeptide of type I collagen (â-CTX) and association with response and progression.
4. To describe overall response rate (proportion of participants who achieve a best response of complete response or partial response using RECIST 1.1 criteria), time until progression (time from initiation of systemic treatment to the date of documented disease progression), and progression-free survival (time between the first date of systemic treatment to first date of documented progression or death due to any cause).
5. To describe incidence of skeletal related events defined as a composite of pathologic fracture, spinal cord compression, radiation or surgery to bone, and hypercalcemia of malignancy.

2.3 Exploratory Objective:

1. OPTIONAL: To describe findings in Extreme CT scan at baseline and/or at 6 months and association with skeletal related events.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, the subject must meet all of the inclusion and none of the exclusion criteria.

1. Signed Written Informed Consent
2. Ability to understand and the willingness to sign a written informed consent document.
3. Participants must have signed and dated an IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal participant care.
4. Participants must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and serial biopsy schedule.
5. Participants must be willing to consent to PA-17-0577, a protocol led by Dr. Jianjun Gao, that allows for tissue sample collection and analysis
6. Type of Participant and Target Disease Characteristics
7. Histological confirmation of RCC with a clear-cell component, including participants who may also have sarcomatoid or rhabdoid features
8. Advanced (not amenable to curative surgery or radiation therapy) or metastatic (AJCC Stage IV) RCC
9. No prior systemic therapy with nivolumab or cabozantinib or previous systemic treatment for metastatic disease.

   ECOG performance status ≤2 (Karnofsky ≥60%) (See Tables 1 and 2 in section 14 for reference)
10. Presence of both a bone metastasis and visceral or soft tissue metastatic lesion amenable to biopsies
11. Patients must have adequate organ and marrow function as defined below:

    * absolute neutrophil count ≥1,000/mcL
    * platelets ≥100,000/mcL
    * total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (Except participants with Gilbert Syndrome who must have a total bilirubin < 3.0 x ULN)
    * AST(SGOT)/ALT(SGPT) ≤3 × institutional ULN
    * GFR ≥30 mL/min (using the Cockcroft-Gault formula)
12. For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
13. Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
14. Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression. Treated CNS metastases are defined as having no ongoing requirement for corticosteroids for at least 2 weeks prior to enrollment and no evidence of progression or hemorrhage after treatment completed at least 4 weeks prior to enrollment clinical examination and brain imaging (MRI or CT).
15. Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.
16. Patients are eligible to receive standard of care nivolumab and cabozantinib treatment and must be prescribed this regimen at treating physician's determination.
17. Age and Reproductive Status
18. Males and females aged 18 years or greater. Because there is inadequate dosing or adverse event data in patients <18 years of age, children are excluded from this study.
19. The effects of cabozantinib and nivolumab on the developing human fetus are unknown. For this reason and because tyrosine kinase inhibitors and immune checkpoint inhibitors as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation (refer to MDA Policy CLN 1114) and for 4 months after the last dose of cabozantinib and 4 months after the last dose of nivolumab. This includes all female patients, between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following:

    Postmenopausal (no menses in greater than or equal to 12 consecutive months).
    * History of hysterectomy or bilateral salpingo-oophorectomy
    * Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
    * History of bilateral tubal ligation or another surgical sterilization procedure.
    * In addition, females < 55 years-of-age must have a serum follicle stimulating (FSH) level > 40 mIU/mL to confirm menopause).
20. Approved methods of birth control are as follows: Hormonal contraception (i.e., birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
21. Males who are sexually active with women of childbearing potential (WOCBP) must agree to follow instructions for method(s) of contraception for the duration of study treatment and 7 months after the last dose of study treatment (ie, 90 days [duration of sperm turnover] plus the time required for the investigational drug to undergo approximately five half-lives).
22. Azoospermic males are exempt from contraceptive requirements. WOCBP who are continuously not heterosexually active are also exempt from contraceptive requirements, and still must undergo pregnancy testing as described in this section. Investigators shall counsel WOCBP, and male participants who are sexually active with WOCBP, on the importance of pregnancy prevention and the implications of an unexpected pregnancy. Investigators shall advise on the use of highly effective methods of contraception which have a failure rate of < 1% when used consistently and correctly.

Exclusion Criteria:

Any active CNS metastases greater than 0.5cm in size. Participants with treated CNS metastases demonstrated stability for at least 28 days are allowed to enroll.

1. Any impending pathologic fracture or cord compression requiring urgent surgical or site-directed therapy. Participants may be eligible if they undergo initial surgery with tissue collection and have adequately recovered and have received clearance for systemic treatment from orthopedic surgeon or neurosurgery. The tissue collected at the time of initial surgery may be used as the baseline tissue collection. An alternative bone metastasis must be available for biopsy after treatment to be considered eligible.
2. Any active, known or suspected autoimmune disease. Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.

   Any condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of enrollment. Inhaled or topical steroids, and adrenal replacement steroid doses ≤ 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease. Transient short-term use of systemic corticosteroids for allergic conditions (e.g., contrast allergy) is also allowed.
3. Any tumor invading the GI tract or any evidence of endotracheal or endobronchial tumor within 30 days prior to randomization
4. Known history of positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS). Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
5. Known medical condition (e.g., a condition associated with diarrhea or acute diverticulitis, aortic aneurysm, aortic dissection) that, in the investigator's opinion, would increase the risk associated with study participation or study drug administration or interfere with the interpretation of safety results
6. History of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess, bowel obstruction, or gastric outlet obstruction within the past 6 months prior to enrollment
7. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of cabozantinib (e.g., malabsorptive disorder, ulcerative disease, uncontrolled nausea, vomiting, diarrhea, or small bowel resection)
8. Serious, non-healing wound or ulcer within 2 weeks prior to study enrollment. May be eligible if cleared by surgical team.
9. Evidence of active bleeding or bleeding susceptibility; or medically significant hemorrhage within prior 3 months prior to study enrollment. Microscopic hematuria is allowed.
10. History of cerebrovascular accident (CVA) including transient ischemic attack within the last 6 months prior to enrollment unstable cardiac arrhythmia within 6 months prior to enrollment
11. Prolongation of the Fridericia corrected QT (QTcF) interval defined as > 450 msec for males and > 470 msec for females, where QTcF = QT / 3√RR with triplicate measurements
12. Poorly controlled hypertension (defined as systolic blood pressure (SBP) of > 150 mmHg or diastolic blood pressure (DBP) of > 90 mmHg), despite antihypertensive therapy
13. History of any of the following cardiovascular conditions within 3 months of study enrollment: cardiac angioplasty or stenting, myocardial infarction, unstable angina, coronary artery by-pass graft surgery, symptomatic peripheral vascular disease, class III or IV congestive heart failure (CHF), as defined by the New York Heart Association (NYHA)
14. Any radiologic or clinical evidence of pancreatitis within 30 days prior to enrollment
15. Inability to swallow oral medications or unwillingness or inability to receive IV administration.

    History of allergic reactions attributed to compounds of similar chemical or biologic composition to cabozantinib or other agents used in study.
16. Pregnant women are excluded from this because cabozantinib is a class D agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with cabozantinib breastfeeding should be discontinued if the mother is treated with cabozantinib. The potential risks may also apply to other agents used in this study.
17. Administration of a live, attenuated vaccine within 30 days before first dose of study treatment.
18. Active infection requiring systemic treatment. Acute or chronic hepatitis B or C infection or known positive test for tuberculosis infection where there is clinical or radiographic evidence of active mycobacterial infection.
19. History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
20. Prior/Concomitant Therapy
21. Prior treatment with cabozantinib
22. Concomitant strong CYP3A4 inducers or inhibitors (e.g., dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbital, and St. John's Wort).
23. Concomitant treatment, in therapeutic doses, with warfarin or warfarin-related agents, direct thrombin inhibitors (e.g., dabigatran), direct factor Xa inhibitor betrixaban, or platelet inhibitors (e.g., clopidogrel). Allowed anticoagulants are the following:
24. Prophylactic use of low-dose aspirin for cardio-protection (per local applicable guidelines) and low-dose low molecular weight heparins (LMWH).
25. Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in subjects without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor.
26. Major surgery (e.g., nephrectomy, laminectomy, open pedicle screw stabilization) less than 4 weeks prior to study enrollment. Procedures not classified as major surgery: percutaneous stabilization, kyphoplasty, and laser interstitial thermal therapy (LITT) and can enroll on study 1-2 weeks after procedure.
27. Physical and Laboratory Test Findings
28. WBC < 2000/μL
29. Neutrophils < 1500/μL
30. Platelets < 100 x 103/μL
31. Hemoglobin < 9.0 g/dL (support with transfusion is acceptable)
32. Calculated creatinine clearance < 20 mL/min (using the Cockcroft-Gault formula)
33. AST/ALT > 3.0 x ULN
34. Total bilirubin > 1.5 x ULN (except participants with Gilbert Syndrome who must have a total bilirubin level of < 3.0 x ULN)
35. Urine protein/creatinine ratio (UPCR) ≥ 1.0, unless 24-hour urine protein is < 1.0 g
36. INR > 1.6
37. History of allergy or hypersensitivity to study drug components
38. History of severe hypersensitivity to a monoclonal antibody
39. Other Exclusion Criteria
40. Prisoners or participants who are involuntarily incarcerated.
41. Participants who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2027-04-07 (Estimated); Study Completion 2029-04-07 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Campbell, MD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org